CLINICAL TRIAL: NCT06610695
Title: Advanced Molecular Imaging of Cholestatic Disorders in Humans: Pathophysiological Characterization
Brief Title: PET/CT Scans Using the Tracer 11C-Csar, a Bile Acid Analog, to Depict and Visualize Cholestatic Disorders in Patients with Genetic Liver Disorders and Healthy Individuals
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Csar_Cholestatic and healthy; 1-10-72-203-23 (Other: The Central Denmark Region Committees on Health Research Ethic)
Record Dates: First submitted 2024-08-30; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Cholestasis; Genetic Liver Disorder
Keywords: cholestasis
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Bloodsamples for a biobank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Purpose The primary goal is to study liver diseases with defects in bile excretion. Investigators aim to do this using a radioactive tracer that mimics human bile and can be visualized with a PET/CT scanner. This will help us understand where these defects occur and how they might be treated in the future.

Background Patients with liver diseases affecting bile excretion are at risk of developing cirrhosis. When bile cannot be excreted normally, it accumulates in the liver, damaging its function. It can also build up in the skin, causing yellowing and itching. Currently, patients are monitored using blood tests that do not always reflect the severity of liver disease. There are a few medications available, but they have limited efficacy.

Advanced PET/CT scanning with the radioactive tracer 11C-Csar offers a way to investigate this. 11C-Csar has been developed, tested, and approved for human use at Aarhus University Hospital and has been used in previous patient studies.

The study aims to use this method to show how 11C-Csar moves through the liver and bile ducts in both healthy individuals and patients with a genetic liver disease. Investigators aim to:

* Observe how defects affect the liver handling of bile acids.
* Determine the excretion kinetics of 11C-Csar, including specific rate constants.
* Compare standard blood tests with 11C-Csar PET/CT findings to assess how well blood tests reflect actual liver damage.
* Visualize potential targets for future interventions.

Study Plan The scientific study involves a single examination day at the Department of Nuclear Medicine and PET. Participants will arrive fasting in the morning. An intravenous line will be placed in both arm veins, a catheter in a wrist vessel, and a hepatic vein catheter. The hepatic vein catheter will be inserted by a trained liver specialist using local anesthesia and ultrasound guidance, confirmed by X-ray. The tracer 11C-Csar and the dye indocyanine green (ICG) will be administered through the IV lines. ICG will be infused 90 minutes before scanning, and 11C-Csar will be administered at the start of the scan. Blood samples will be taken from the liver and wrist during the scan, which lasts about 45 minutes. After the scan, the catheters will be removed, and the participant can go home shortly after. Approximately 250-300 ml of blood will be drawn, which poses no risk to the participants. The total participation time is expected to be around 4 hours. Some patients may be offered a second scan if they develop new symptoms, repeating the scan when liver blood tests normalize.

Participants Patients with bile accumulation liver diseases will be informed of the study during visits to the Department of Hepatology and Gastroenterology, AUH. Healthy controls will be recruited through advertisements on webpages dedicated for the purpuse. Interested individuals will receive written information.

Side Effects, Risks, and Discomfort The risk of phlebitis and bleeding from IV insertion is minimal, as these procedures are performed daily.

The total radiation exposure from the PET/CT scan with 11C-Csar is 2.5 mSv.

Funding The study is researcher-initiated, with no financial interests for the involved researchers.

Publication of Results Both negative, positive, and inconclusive results will be published. The study results will be submitted to peer-reviewed international journals in liver disease and/or radiology and presented at national and international scientific conferences.

Ethics The study will be conducted following the principles of the Helsinki Declaration II with amendments and after approval by the Regional Ethics Committee for Midtjylland. While there is no immediate benefit for patients, the results will enhance our understanding of liver disease with bile acid accumulation. Investigators believe the risks and potential side effects are outweighed by the expected benefits.

DETAILED DESCRIPTION:
Background

Cholestasis is defined as a decreased flow of bile from the liver to the duodenum, either due to reduced excretion from the liver, defects in the enterohepatic circulation or blockage of the biliary tree. Bile acids are essential for the absorption of lipophilic compounds from the intestine. [1] When bile acids accumulate in the liver, it causes damage to the tissue.

Patients with cholestasis typically present with jaundice and pruritus caused by the bile acids accumulating in the skin. Elevated blood levels of alkaline phosphatases (AP), gamma-glutamyl transferase, and sometimes bilirubin are observed [2]. The clinical workup includes ultrasound sonography (US) to exclude tumours/stones and specific blood tests, including autoantibodies, immunoglobulins, etc. A thorough history of familial diseases and medicine intake is also important for workup [1]. A liver biopsy can be necessary to evaluate hepatic histopathological changes in the liver. Treatment depends on the specific cause. The present project deals with medical causes of cholestasis as described below, i.e., not mechanical obstruction such as cancer or gallstones.

Monitoring medical cholestatic disorders relies on continuous blood measurements of AP, bilirubin, etc. Still, these tests do not necessarily convey information about the degree of cholestasis from a functional point of view.

The enterohepatic circulation Intact enterohepatic circulation is important since de novo synthesis of bile acids does not play a significant role in enterohepatic circulation.[3] Bile acids are absorbed in the terminal ilium by the ileal bile acid transporter (ASBT/SLC10A2) and secreted into the portal vein, which delivers the bile acids back to the liver. Here, the Na+-taurocholate co-transporting peptide (NTCP) and organic anion- transporting proteins (OATPs) mediate bile uptake from the sinusoids to hepatocytes.[4] The bile salt export pump (BSEP) facilitates the transport from hepatocytes into bile canaliculi. The multidrug resistance proteins 3 and 4 (MRP3/ABCC3, MRP4/ABCC4) and the heteromeric organic solute transporter (OSTa/b/SLC51A/SLC51B) mediate backflux from hepatocytes to blood. [3] All these transporters can be defective in different genetic diseases and lead to cholestasis, which is the case in patients with progressive familial intrahepatic cholestasis (PFIC), including protein-truncating mutations in tight-junction protein 2 gene (TJP2) and mutations in bile salt export pump (BSEP). Some of these patients will debut with drug-induced liver disease (DILI) or have recurrent cholestasis.

The functional consequences of genetic mutations and variations affecting hepatic transporter and tight- junction proteins as the cause of cholestatic disorders have been challenging to study in vivo. Some disorders progress rapidly into cirrhosis and potentially hepatocellular carcinomas, whereas others do not become apparent until the partially defective transporter protein is as it can be seen in drug-induced liver injury (DILI), e.g., for substrates excreted into bile via bile salt exporting protein, BSEP [5]-[9] Studying the hepatobiliary handling of bile acids has been challenging, primarily due to the livers concealed position between the portal venous and systemic blood systems and because of the inherent difficulty in retrieving sampling materials from bile.

In the present project, investigators wish to generate novel insights into the functional effects of cholestasis by visualizing the handling of bile acids. Visualization is achieved by using functional positron emission tomography/computer tomography (PET/CT).

Previous studies The Department of Hepatology & Gastroenterology and the Department of Nuclear Medicine & PET Centre, both Aarhus University Hospital, have, in collaboration, developed a PET/CT method to study the enterohepatic circulation of bile acids. This method utilizes the carbon-11 labelled conjugated bile acid tracer cholylsarcosine (11C-CSAR) [3], [10]-[12].

11C-CSAR is a synthetic conjugate of N-methyl glycine (sarcosine) and cholic acid, which was chosen due to its similarity to taurocholic acid, one of the essential bile salts in humans. Also, this bile acid is not metabolized in the body or by bacteria in the intestines.

Investigators have validated the 11C-CSAR PET/CT method in patients with various cholestatic disorders and healthy controls. [3], [11]-[14] Investigators plan to expand our data pool using newer and more advanced scanners and to expand the method to patients with genetic mutations/variations in proteins involved in biliary secretion to learn about these conditions and functional effects. Examination of this patient group has not been done before.

Hypothesis

* The hepatobiliary secretion of 11C-Csar will be reduced in patients compared to healthy individuals.
* Cholestatic disorders affect different steps in hepatobiliary secretion of bile acids from blood depending on the specific disease/genetic disorder
* The functional effect of cholestatic disorders varies among patients with some patients being almost unaffected and others being severely affected.
* The measurements from functional11C-CSar PET/CT provide a better evaluation/description/characterization of patients with cholestatic disorders than standard biochemistry.

Study design The study is an investigator-initiated observational study. Healthy volunteers, patients who present with cholestasis and patients with known genetic disorders in the hepatobiliary system will be offered participation in a functional 11C-CSAR PET/CT.

Participants arrive at the department at 8.00 AM after an overnight fast. The participants will get a hepatic vein catheter, two venous catheters and an artflon. Indocyanine green (ICG) will be administered intravenously to measure hepatic flow (Ficks principle).

11C-CSAR is administered intravenously at the beginning of a functional PET/CT. The PET/CT scan takes approximately 45 minutes. Blood samples will be drawn from the artflon and the hepatic vein catheter during the scan to measure the hepatic blood flow and the concentrations of 11C-CSAR.

Investigators aim to include 14 patients with different cholestatic disorders, including genetic disorders, and eight healthy volunteers.

Methods 11C-CSAR PET/CT 11C-CSAR is injected intravenously in micro-doses and enters the enterohepatic circulation of endogenous bile acids [3], [10]-[13]. The tracer is injected at the beginning of a dynamic PET/CT scan of the hepato-biliary system. By external detection, this method provides real-time measurements of the time course of tissue concentrations of 11C-CSAR in liver tissue, bile ducts, etc. Combined with arterial blood measurements from an artflon and hepatic blood flow measurements using ICG (Ficks principle), specific kinetic parameters of the livers handling of conjugated bile acids are calculated by fitting a mathematical model to data. These parameters include uptake from sinusoidal blood, back flux to sinusoids, transport from hepatocytes into biliary canaliculi, and bile flow. Mean transit time in hepatocyte and relative tissue concentrations are also calculated [3], [10]-[13].

The 11C-CSAR PET/CT scans will be performed after an overnight (8-hour) fast, and the participants cannot take their regular medication before the scan. The participants will be placed in a supine position in the Siemens Biograph Vision Quadra with the liver within the 106 cm field of view. A low-dose CT scan is performed to visualize the anatomy. 50 MBq 11C-Csar mixed in 10 ml of saline water is administered intravenously over 25 seconds at the beginning of a 45-minute functional 11C-CSAR PET/CT scan. During the scan, blood samples from the hepatic vein catheter are collected to measure concentrations of 11C-CSAR.

Tracer The 11C-CSAR tracer will be prepared at the Department of Nuclear Medicine and PET Centre, Aarhus University Hospital, using a 3-step radio-synthesis method. [16]

Preparation Patients with cholestasis are followed with blood samples in the departments. Before the scan of the volunteers, blood samples are taken for biochemical analysis (haemoglobin, leukocytes, thrombocytes, INR, CRP, alanine transferase, bilirubin, alkaline phosphatase, creatinine, eGFR, albumin, sodium, potassium, and possibly other relevant health-related parameters), to rule out unknown health issues related to the liver. The amount of blood is 20 ml, which will be drawn at the time of inclusion at the Department of Clinical Biochemistry or by us. The results of the blood samples will appear in the participants regular medical journals. The blood samples are discarded immediately after analysis.

Women participating in the study will be asked to take a pregnancy test on the day of the scan. The test will be performed on urine. The urine will be discarded afterwards.

Catheters Venflons are placed percutaneously in both cubital veins by a trained technician for intravenous administrations of 11C-CSAR and ICG. For blood sampling, an artflon catheter will be placed percutaneously in a radial artery by a trained anesthesiologist, and a catheter will be placed in the hepatic vein via the right jugular vein by a trained hepatologist.

Data assessment The PET data involves 11C-CSAR concentrations in liver and bile ducts and blood concentrations of 11C-CSAR in arterial and hepatic vein blood and hepatic blood flow. Investigators will calculate the kinetics of hepatobiliary excretion of 11C-CSAR from the patients with cholestasis and compare them with the healthy volunteers.

Data management Source data for each participant is registered in the participants PET journal or Case Report Form (CRF). The CRF is established as a project in REDCap and contains information on contact information and demography (sex, weight, height). Source data on blood work will be in Labka, EPJ (Electronic patient journal).

The PET journal contains all data considering tracer production, quality control, administered dose, and scan data (including side effects related to the scan). The localization of source data is kept in the trial master file (TMF). The signed consent forms are kept in digital form in REDCap, and a physical form is kept in a locker with the TMF. Data is held in the eCRF (REDCap) and the PET journal.

Source data on each participant includes all data regarding the production of tracer and quality control, administered dose, data on scan results and possible deviations and complications, as well as the participants health records and laboratory results. This data will be registered in each participants PET journal and CRF.

All research participants will perform data management and assessment. Sample sizes and statistics The number of healthy subjects (n=8) is based on our experience from previous PET studies, including 11C-CSar studies.

The patient group is expected to be very heterogeneous, with individual results ranging from numbers close to healthy subjects to values significantly different from healthy subjects. As there are only so many patients with genetic disorders, Investigators aim to include 14 during the period to get a broad range of patients.

The statistical analysis is carried out in STATA and GraphPad Prism in pseudonymized form. Data is deleted or anonymized after ten years.

Data will be analyzed per protocol and participants who lack data considering the primary endpoints will be excluded from the analysis. It will be stated in the results if any deviations from the statistical analysis plan occur. Should a participant withdraw from the study before completion, a new participant will be recruited to ensure to have a complete dataset of participants.

Risk, side effects and precautions Monitoring during 11C-CSAR PET/CT During 11C-CSAR PET/CT, participants will be under constant medical supervision. The Department of Nuclear Medicine and PET Centre has all the necessary equipment and medication in case of acute tracer-related reactions. The personnel monitoring the participants are trained in treating critical allergic responses. No allergic reactions is anticipated as the tracer 11C-CSAR acts like taurocholic acid, which is an endogenous bile salt in humans. The ICG poses a minimal risk of allergic reactions. Any reactions will be monitored closely and reacted upon.

Radiation risk The amount of tracer, 11C-Csar, will depend on the patient weight: 0,5 MBq/kg body weight will be administered, with a minimum level of 25 MBq and a maximum of 50 MBq. Former studies have shown that 11C-Csar performs a radiation risk of 0,0062 mSv/MBq[15]. Therefore, an average person weighing 75 kg will have a radiation exposure of 0,23 mSv. The radiation dose from the low-dose CT scan is 2,3 mSv. The radiation exposure if a patient is scanned once is 2,5 mSv. Few of our patients will be offered a second scan, resulting in a total radiation exposure of 5 mSv.

As per appendix II: Use of Ionizing Radiation in Health Science Research "(Retningslinjer om anvendelse af ioniserende stråling i sundhedsvidenskabelige forsøg)" this corresponds to the risk category IIb. Compared to the annual background radiation, which is 3 mSv, the given value of 2,5 - 5 mSv represents a relatively small contribution.

A total dose of 5 mSv can be calculated to increase lifetime cancer risk by 0.025% due to participation in this study. This is relative to the normal 25% lifetime cancer risk.

Side effects 11C-CSAR is a synthetic conjugate of N-methyl glycine (sarcosine) and cholic acid, which was chosen due to its similarity to taurocholic acid, one of humans most essential bile salts. No side effects have previously been seen or are expected.

ICG is used as a routine test for measuring hepatic flow, and adverse events are infrequent.

Catheters The participants will have venous catheters placed in each cubital vein, an artflon in the radial artery, and a hepatic vein catheter via the right jugular vein. Insertion of the catheters may cause a small amount of pain, subcutaneous bleeding and pose a minimal risk of superficial infection. These catheters are used daily in the hospital without any side effects.

Blood samples During the 11C-CSAR PET/CT scan, blood samples from the participants will be drawn from the artflon in the radial artery and the hepatic vein catheter. In total, 250 - 300 ml of blood will be drawn from the participants. This blood loss is of no risk for the participants, and the blood will be discarded immediately after analysis.

Monitoring after the trial All catheters are removed after the 11C-CSAR PET/CT scan, and the participants can go home 30 minutes after the scan.

All participants will be encouraged to contact us if they feel discomfort or have concerns regarding the trial and the scans after participating.

Information from medical records The investigator will receive pass-on information from the electronic medical records (Midt-EPJ) regarding patients listed on the outpatient lists and admission in the bed wards (fulfilment of in- and exclusion criteria) prior to obtaining informed consent, and the information will be passed on to the project afterwards. Before obtaining informed consent, information from about 50 patients will be passed on to the investigator. This information is based on records from the past five years. Information from the participating patients medical charts will be collected for the project from all 14 patients after obtaining written, informed consent. The informed consent gives the investigator and the investigator representatives direct access to information about the study participants; health status from their electronic medical patient records. The data include, gender, age, medical history, current medication, biopsy results, pathology reports and biochemical test results. The consent provides the investigators, their representatives, and any regulatory authority direct access to obtain information from the patients medical records, including electronic records, for the purpose of reviewing the study participants health status necessary for the implementation of the research project and for monitoring purposes, including self-inspection, quality control, and monitoring, which they are obligated to perform.

Respect for the physical and mental integrity and the privacy of the study participants The study will be registered in the Region Midt study register. All data will be treated confidentially and according to the applicable Danish legislation.

When participants have signed a consent, information from their health records will be collected, according to §43, 1 in the Danish Health Law.

The data will be utilized in the scientific publication of the study findings and will undergo complete anonymization, ensuring that no personally identifiable information is disclosed. Information regarding the participants will be protected according to the General Data Protection Regulation (GDPR), the Data Protection Act, and the Danish Health Law §43 will be complied with.

Financial statement The involved scientists initiated the study, and none of the involved partners have any economic interests in the study. The project is financed by Novo Nordisk Fonden (1 million DKK, part of a grant totaling 8.506500,00 million DKK). The grants are provided for a more extensive research program on liver disease and imaging modalities (given to Michael Sørensen). The expenses include the salary for PhD student Maja Kanstrup Jørgensen and all expenses regarding the study, including but not limited to scans, blood samples, and compensation to the participants. Regnskabsafdelingen, AUH, administers the amount.

Reimbursement The patients will not receive reimbursement, but travel expenses, overnight stays at the patients hotel if necessary, and documented lost wages will be covered.

Healthy participants are offered 1500 DKK for participation in addition to documented travel expenses and lost wages. Participants must pay taxes on the specified amount, and reimbursement for the study participant will only be provided after the scheduled scanning day. If the healthy participants withdraw from the study before the scheduled scan, no reimbursement will be provided.

Eligible patients are identified from the outpatient and admission lists of the bed wards at the Department of Hepatology and Gastroenterology, Aarhus University Hospital, and the Department of Internal Medicine, Regional Hospital of Viborg.

If the patient shows interest in the project, Maja or Michael will give oral information about the project. If the patient is still interested, the written project information and the brochure: Research Participants' Rights in a Health Science Research Project" will be handed out or sent via E-boks.

When the person has read the material, the primary investigator, Maja, will have an in-depth discussion with the participant about the nature of the study and the rights of the trial subject. Participant will be informed about the right to bring an assessor, the right to consider for up to 24 hours, and how they can withdraw their consent at any time without reason. The conversation will occur in quiet surroundings with enough time to discuss the study thoroughly. The investigator will ensure that the participant understands the matter of the investigation.

Written and verbally informed consent will be obtained before participation in the study can begin. Information about the possibilities of complaint and possible compensation regarding unforeseen side effects is given.

Healthy individuals The healthy individuals will be recruited through internet advertisements on the Facebook group "Forsøgspersoner Aarhus Universitet" and the webpages forsøgspersoner.dk, forskning.nu.

Interested healthy individuals will be encouraged to contact the primary investigator, Maja. A meeting will be arranged to give oral information on the project in the same way as mentioned in the previous section. Routine blood samples will be drawn to ensure no liver disease is present.

The 11C-CSAR PET/CT scan is booked when a signed consent is made.

Publication of the results All positive, negative, or inconclusive results will be published. Results will be presented at Danish and international meetings and published in international peer-reviewed scientific journals with author lists according to the ICMJE recommendations.

Ethical aspects of the study The tests are carried out under the principles of the Helsinki Declaration II with appendix after approval by The Committee on Health Research Ethics for Region Midt. Inclusion of participants follows the ethical guidelines set out by The Ethics Committee on request upon participation, obtainment of informed consent, information on trial subjects rights, etc.

11C-CSAR PET/CT has been used several times in patients and healthy individuals in the department without any adverse events. As mentioned, the tracer 11C-CSAR has no therapeutical effect and is quickly removed from the body.

ICG is often used clinically to measure hepatic flow, and adverse events are infrequent.

There is no direct benefit for the participants, but the results will hopefully increase our insight in patients with cholestasis. Patients will not experience any delay in their regular treatment.

In our opinion, the risks and possible side effects are outweighed by the expected benefits.

When signing the informed consent letter, participants will decide if they want information on unexpected findings in the scans. Should incidental results occur during the scans, the participants will be informed and offered regular clinical examinations.

Criteria for interruption of the study for each patient

* The participant withdraws the consent.
* The responsible physician considers the participants health endangered by continuing the trial. Criteria for interruption of the study
* Unexpected severe adverse events related to the trial in more than one participant.

Insurance Patienterstatningen; will cover subjects if necessary. Timeline Inclusion will start shortly after approval from The Committee on Health Research Ethics for Region Midt. PET/CT scans will be planned weekly when the patients are in the departments. The project is terminated after the last scan is completed or no later than five years after the approval of the study. Investigators will perform data management concurrently and finish it within the duration of the PhD project.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion of healthy individuals
* No prior or current history of liver diseases
* No medication that interferes with the hepatobiliary system
* Age above 18
* A signed consent must be present on the day of the 11-CSAR PET/CT scan.
* A negative pregnancy test performed on the day of the scan.

Exclusion Criteria:

* Prior cholecystectomy
* Pregnancy
* Assessed ineligibility by a medical doctor based on blood parameters measured at inclusion if these are abnormal.
* Claustrophobia or the inability to remain still during a 45-minute scan.

Criteria for inclusion of patients with cholestasis

* Cholestasis at the time of inclusion, measured by elevated AP, bilirubin, or both.
* Ultrasound sonography which ruled out mechanical obstruction.
* Age above 18
* A signed consent must be present on the day of the 11C-CSAR PET/CT scan.
* A negative pregnancy test performed on the day of the scan. Criteria for exclusion of patients with cholestasis
* Pregnancy
* Claustrophobia or the inability to remain still during a 45-minute scan.
* Coagulation deficiency that does not allow hepatic vein catheter (relative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects We plan to include eight healthy individuals and 14 patients with different cholestatic disorders.
  We aim to include patients with different genetic disorders affecting the hepatobiliary transport of bile acids. This includes, but is not limited to, patients with progressive familial intrahepatic cholestasis (PFIC), including protein-truncating mutations in tight-junction protein 2 gene (TJP2) and mutations in bile salt export pump (BSEP).
  The healthy individuals will be recruited through internet advertisements on the Facebook group "Forsøgspersoner Aarhus Universitet" and the webpages forsøgspersoner.dk, forskning.nu.
  Interested healthy individuals will be encouraged to contact the primary investigator, Maja. A meeting will be arranged to give oral information on the project in the same way as mentioned in the previous section. Routine blood samples will be drawn to ensure no liver disease is present.
  The 11C-CSAR PET/CT scan is booked when a signed consent is made.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to apply the 11C-CSAR PET/CT method to quantify hepatobiliary secretion kinetics of 11C-Csar in both healthy human participants and patients with various cholestatic disorders, including those of genetic origin. | through study completion, an average of 2 years
  Changes in the hepatobiliary excretion kinetics of 11C-CSar between patients and healthy

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Hepatology and Gastroeneterology Aarhus University Hospital., Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided